CLINICAL TRIAL: NCT00434005
Title: Effect of Diesel Exhaust Particulate Exposures on Endothelial Function in Humans - the Role of Oxidative Stress
Brief Title: Effect of Diesel Exhaust Particulate Exposures on Endothelial Function in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Joel Daniel Kaufman, Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 22969-D; R830954; R827355; MO1RR-00037; ES015915; ES013195
Record Dates: First submitted 2006-08-25; First posted 2007-02-12 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Air pollution; diesel; antioxidant; oxidative stress; endothelial; HRV; BAR
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diesel Exhaust (Experimental)
  Interventions: Drug: N-acetylcysteine, ascorbate; Drug: Placebo
- Filtered Air (Sham Comparator)
  Interventions: Drug: N-acetylcysteine, ascorbate; Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine, ascorbate — NAC: 600mg twice daily for the day prior to exposure and 1x pre-exposure Ascorbate: 500mg twice daily for 7 days prior to exposure
Drug: Placebo — matched appearance to acetylcysteine and ascorbate intervention

SUMMARY:
Objectives: This proposal addresses the overall hypothesis that ambient fine particulate matter exerts cardiovascular health effects via alteration of endothelial homeostasis, through a mechanism mediated by oxidative stress. This project will use a controlled human inhalation exposure to diesel exhaust particulate (DEP) as a model to address the following objectives: 1) Determine whether exposure to inhaled DEP is associated with endothelial dysfunction in a concentration-related manner; 2) Determine whether exposure to inhaled DEP is associated with evidence of systemic oxidative stress; and 3) Determine whether antioxidant supplementation blunts the DEP effect on endothelial function.

DETAILED DESCRIPTION:
OBJECTIVES Evidence of the cardiovascular health effects of both acute and chronic exposure to ambient fine particulate matter (PM) has continued to accumulate in epidemiologic and experimental studies, without a demonstrated coherent pathophysiologic explanation. At the same time, the role of endothelial homeostasis in the development and triggering of cardiovascular disease has become more clear and compelling. Importantly, oxidative stress has emerged as a potential link between these two developments: Oxidative stress is known to play a role in endothelial dysfunction and is exerted by components of PM, especially of PM from combustion products. Based on this we propose an overall hypothesis: Inhalation of combustion-derived particles impact cardiovascular health by impairing endothelial function, through mechanisms mediated by increased oxidative stress.

Diesel exhaust particulate (DEP), an important contributor to ambient fine PM, has been demonstrated to exert oxidative stress in experimental systems. We propose a series of experiments to explore whether human exposure to DEP results in alteration of endothelial homeostasis and evidence of oxidative stress, and whether an antioxidant regimen can blunt the effects on endothelial function.

The objectives of this proposed research are to address the following specific hypotheses:

1. Human exposure to inhaled DEP (at concentrations approximating 0, 100, 200 μg PM2.5/m3 [PM less than 2.5 microns in aerodynamic diameter]) results in concentration-related alteration of endothelial homeostasis, as reflected in ultrasonographic measurement of the brachial artery, plasma markers of endothelial homeostasis (endothelin-1, ICAM-1 [intercellular adhesion molecule-1], e-selectin, nitric oxide metabolites nitrate [NO3-] and nitrite [NO2-], IL-6, and TNF-α), and markers of thrombosis associated with endothelial activation or injury (plasminogen activator inhibitor-1 [PAI-1], Von Willebrand's factor [VWF], and D-dimer).
2. Human exposure to inhaled DEP at 200 µg PM2.5/m3 results in evidence of systemic oxidative stress as assessed by markers in plasma and urine (isoprostane F-2α).
3. Reduction in oxidant stress by ascorbate and N-acetylcysteine supplementation blunts the effect of inhaled DEP on endothelial function, as determined by ultrasonographic assessment of the brachial artery, plasma markers of endothelial homeostasis, or markers of thrombosis associated with endothelial activation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-49.

Exclusion Criteria:

* Nonsmokers, no history of hypertension, asthma, diabetes, hypercholesterolemia, or other chronic conditions requiring ongoing medical care. No recent history of antioxidant, vitamin/mineral/botanical, or fatty acid supplementation beyond a daily multi-vitamin.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Brachial artery caliber | Pre-exposure, immediate post-exposure

SECONDARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation | Post-Exposure
Plasma Endothelin-1 | Post-exposure (adjusted for pre-exposure level)
Serum IL-6 | Post-exposure (adjusted for pre-exposure level)

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Kaufman, M.D., MPH, Principal Investigator — University of Washington
Locations (1):
- Northlake Laboratory, Seattle, Washington, United States

REFERENCES:
- [Derived] Cosselman KE, Krishnan RM, Oron AP, Jansen K, Peretz A, Sullivan JH, Larson TV, Kaufman JD. Blood pressure response to controlled diesel exhaust exposure in human subjects. Hypertension. 2012 May;59(5):943-8. doi: 10.1161/HYPERTENSIONAHA.111.186593. Epub 2012 Mar 19. PMID 22431582
- See also: Controlled Exposure Laboratory — http://depts.washington.edu/envhlth/nlakeexplab/index.html